CLINICAL TRIAL: NCT05521763
Title: Seasonal Influenza Vaccine Uptake Among Health Care Workers Following Awareness and Availability of Influenza Vaccine Supply in Tertiary Care Hospitals, Bangladesh
Brief Title: Influenza Vaccine Uptake Among Healthcare Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Institute of Epidemiology, Disease Control and Research (Other); Sylhet M.A.G.Osmani Medical College (Other); Mymensingh Medical College Hospital (Unknown); Rajshahi Medical College (Other); Khulna Medical College Hospital (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR-21150
Record Dates: First submitted 2022-08-17; First posted 2022-08-30 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Influenza Vaccines
Keywords: Vaccination Awareness; Healthcare Workers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention package with the availability of vaccine supply only (Experimental): 1. The investigators will work with the supplier to make that vaccine available at the hospital premises. Then a vaccination booth will be set up at the hospital premises and will administer the vaccine at the MRP.
  2. All HCWs will be notified about only vaccine availability information by the hospital director and respective heads.
  3. A list of all staff working in the study hospitals will be prepared, and they will be provided with an influenza vaccination record card with a unique identification number. The study staff will ensure receipt of vaccination cards for all participants.
  4. A short message (SMS) will be delivered over the mobile phone number to all participants, e.g. vaccination program duration, venue, time, vaccine price, to cascade vaccination information to participants.
  5. Posters with only vaccine delivery information (i.e. vaccination duration, vaccination venue, vaccine price) will be displayed at key hospital locations.
  Interventions: Behavioral: ensuring the availability of influenza vaccine supply & developing influenza vaccine awareness
- Intervention package with vaccinationation awareness only (Experimental): 1. The hospital director and respective heads will notify all HCWs about participating in the vaccination awareness program facilitated by the study team.
  2. The investigators will arrange separate seminars for each group of HCWs in the hospital to sensitize participants about the significance of receiving the influenza vaccine and the risk and benefits of influenza vaccination.
  3. Posters containing messages on the importance of influenza vaccination will be displayed at key hospital locations, e.g., the main entrance of the hospital, nursing station, vaccine delivery point/place, doctors' room, nurses' room, intern doctors' room, common room canteen etc.
  Interventions: Behavioral: ensuring the availability of influenza vaccine supply & developing influenza vaccine awareness
- Intervention package with a combination of vaccine availability and awareness (Experimental): 1. The investigators will work with the study hospital authority, Influenza vaccine manufacturer, and supplier company to set up a vaccination booth at the hospital premises to administer the vaccine at the market-rated price (MRP) by hospital nurses.
  2. The hospital director and respective department heads will notify all HCWs to receive the offered influenza vaccine.
  3. A list of all staff working in the study hospitals will be prepared, and they will be provided with an influenza vaccination record card with a unique identification number.
  4. The investigators will arrange separate seminars for each group of HCWs in the hospital to sensitize participants about the significance of receiving the influenza vaccine and the risk and benefits of influenza vaccination.
  5. A short message (SMS) will be delivered over the mobile phone number to all participants.
  6. Posters with key messages will be displayed at key hospital locations,
  Interventions: Behavioral: ensuring the availability of influenza vaccine supply & developing influenza vaccine awareness
- No intervention (No Intervention): In the control facility, we will not intervene in the existing knowledge and practice about influenza vaccination of the HCWs.

INTERVENTIONS:
Behavioral: ensuring the availability of influenza vaccine supply & developing influenza vaccine awareness — The four interventions will be:
  i) ensuring the availability of influenza vaccine supply; ii) developing influenza vaccine awareness; iii) both ensuring influenza vaccine supply and developing influenza vaccine awareness and iv) control arm with no intervention.
  Arms: Intervention package with a combination of vaccine availability and awareness; Intervention package with the availability of vaccine supply only; Intervention package with vaccinationation awareness only

SUMMARY:
Background:

1. Burden: Health-care workers (HCWs), such as doctors, nurses, and support staff involved in direct or indirect patient care, are at increased risk of influenza virus infections. HCWs may also transmit and spread influenza among hospitalized patients and other caregivers. HCWs often (40-83%) work while experiencing influenza-like illness (ILI), increasing the likelihood of influenza transmission to colleagues and patients.
2. Knowledge gap: Despite the World Health Organization recommendation for seasonal influenza vaccination among priority target groups such as health care workers, the low-income country such as Bangladesh lacks a seasonal influenza vaccination policy among this high-risk group, and vaccine uptake remains low.
3. Relevance: This study aims to generate preliminary data on HCWs willingness to get seasonal influenza vaccines following vaccine availability and factors associated with vaccine uptakes. The data from the study will support policymakers to increase awareness and develop influenza vaccination policy among top priority groups such as health care workers.

Hypothesis: The investigators hypothesize that awareness and availability of influenza vaccine supply would increase influenza vaccine uptake among health care workers

Objectives:

1. To assess influenza vaccine uptake among healthcare workers (HCWs) following awareness and availability of influenza vaccine supply in study hospitals
2. To explore HCWs barriers and Motivators for influenza vaccine uptake
3. To understand policy makers' perspectives on the feasibility of influenza vaccination among HCWs and to share with the National Immunization Technical Advisory Group (NITAG) for a policy decision regarding influenza vaccination

Methods:

The study will be conducted at four tertiary-level public teaching hospitals in Bangladesh. The investigators will use a cluster randomized controlled trial design. The intervention will be randomly allocated at the facility level and will include four arms: i) availability of influenza vaccine supply; ii) influenza vaccine awareness; iii) both influenza vaccine supply and influenza vaccine awareness, and iv) control arm with no intervention. The investigators will assess influenza vaccine uptake before and after intervention and between different study arms. The investigators will also explore the barriers and motivators of vaccine uptake using a qualitative approach. To understand the policy makers' perspectives and opinions regarding influenza vaccination among health care workers, the investigators will conduct in-depth interviews.

Outcome measures/variables:

1. The proportion of influenza vaccine uptake among health care workers before and after intervention and between different study arms
2. Different motivators and barriers to influenza vaccine uptake

DETAILED DESCRIPTION:
Background :

Influenza annually affects a considerable portion of the world's population, causing significant health, social, and economic consequences. According to the World Health Organization (WHO) estimates influenza infects around 5-15% of adults globally. A collaborative multinational study in 2018 led by the US Centers for Disease Control and Prevention (CDC) found that between 291,000 and 646,000 people worldwide die from seasonal influenza-related respiratory illnesses each year.

Influenza has been a frequent cause of nosocomial outbreaks. Health care workers (HCWs) are at risk of influenza infection due to occupational exposure. In a systematic review of 26 studies and a meta-analysis of 15 studies found an increased risk of influenza among HCWs with a pooled prevalence rate of 6.3%, whereas it is 5.1% for healthy working adults other than healthcare workers. The attack rate among HCWs ranged from 18% to 24% during reported influenza outbreaks. HCWs may not only acquire but also transmit and spread influenza among hospitalized patients. HCWs often (40-83%) work while experiencing influenza-like illness (ILI), increasing the likelihood of influenza transmission to colleagues and patients.

Influenza vaccines are the most effective way to prevent infection and reduce the severity of the disease. Retrospective studies have shown correlations between increases in influenza vaccination among HCWs and decreases in nosocomial influenza in acute care settings. In 2012, the World Health Organization's Strategic Advisory Group of Experts (SAGE) on immunization recommended influenza vaccination for HCWs. WHO SAGE declared the highest priority risk groups in which healthcare workers are at the top of the list. Most developed countries have national policies on immunization against seasonal influenza; however, only 46% (64/138) of LMICs have one.

Despite the WHO vaccination recommendations and mounting scientific evidence on influenza burden and awareness, vaccination coverage rates remain low in LMICs. Persistently low rates of vaccine uptake among HCWs in most countries remain an international concern. Although a great response is seen after offering numerous measures to improve vaccination, the vaccination rate among health care workers remains insignificant. Several studies focused on vaccine uptake rates and associated factors with influenza vaccine acceptance and rejection have been conducted among HCWs in high-income countries in North America and Europe. Few studies have been conducted in LMICs (around 18 studies in sites such as Egypt, Vietnam, Jordan, Kenya, Sierra Leone, Malaysia, Turkey, Tunisia, Iran, China and Lebanon) on influenza vaccine uptake among HCWs. However, no reports are available, particularly from South Asian regions, including Bangladesh.

Studies have shown that interventions such as educational materials and training sessions (e.g. dissemination of information both oral and written to increase awareness and knowledge of the importance of influenza vaccination, including posters, mass mailings, fliers, newsletters, meetings, lectures, presentations, visits by experts or researchers, and videos), improved access to the vaccine, rewards following vaccination, organized efforts to raise vaccine awareness, reminders to get vaccinated, and the use of lead advocates for vaccination can improve influenza vaccine uptake among healthcare workers. A cluster randomized controlled trial among health care workers of 33 Dutch nursing homes conducted in 2010 demonstrated that implementing education and lead advocates resulted in moderate but significantly higher vaccine uptake in the intervention group (25%) compared to the control group (16%) over one influenza season.

Comprehensive reviews on influenza vaccine uptake among healthcare workers have identified several factors that may influence vaccine uptake. The desire for self-protection and to protect family rather than absolute disease risk or desire to protect patients was found as among the main drivers of influenza vaccine uptake among healthcare workers. On the other hand, concerns regarding the safety of the vaccines, low-risk perception, denial of the social benefit of influenza vaccination, low social pressure, lack of perceived behavioural control, negative attitude toward vaccines, not having been previously vaccinated against influenza, not having previously had influenza, lack of adequate influenza-specific knowledge, and lack of access to vaccination facilities were identified as major barriers for vaccine uptake.

In Bangladesh, the annual incidence of influenza-associated hospitalization was estimated at 4.4-6.7 per 1,000 population, and the estimated annual incidence of influenza in outpatients with ILI was 100-170 per 1,000 population. Therefore, the risk of influenza spreading in Bangladeshi healthcare settings is a concern. Studies on tertiary care facilities in Bangladesh showed that HCWs frequently reported hospital-acquired respiratory illnesses. A 2010 study found that 27% (61/226) of HCWs experienced a respiratory illness during the study period. On average, each illness episode lasted 4.3 days, and HCWs worked 230 (89%) of the 260 days they were ill. Another unpublished study estimated the incidence of HCWs' self-reported ILI was 16.3 per 100-person years (95% CI, 13-20) Of the HCWs consented to collect swabs during ILI episodes, 14% (8/56) were tested positive for influenza (flu-A, n = 5; flu-B, n = 3). HCWs worked during 105 (98%) of 107 respiratory illness episodes and 7 (88%) of 8 influenza episodes, increasing the likelihood of influenza transmission in hospital wards. Moreover, with overcrowded hospitals and a lack of infection control practices, the nosocomial transmission of influenza would likely be amplified during a pandemic scenario. This escalates sickness absenteeism among healthcare workers and reduces the workforce in healthcare facilities.

To protect HCWs and reduce nosocomial influenza transmission in both epidemic and pandemic settings, the promotion of influenza vaccination among HCWs is a priority. HCWs' knowledge, attitudes, and perceptions about influenza and influenza vaccine influence HCWs decisions regarding vaccination. Understanding the barriers and motivation of vaccine uptake is required to tailor local influenza vaccination policies and implementation strategies to facilitate and improve vaccine uptake.

The Ministry of Health and Family Welfare (MoH&FW), the Government of the People's Republic of Bangladesh, provides influenza vaccines free of cost to all pilgrims, which is mandatory for Hajj pilgrims from any corner of the world recommended by the Health Ministry of Saudi Arabia. Currently, there is no national influenza vaccination policy available for high-priority risk groups recommended by WHO, such as healthcare workers. At present, influenza vaccines are only available in the private sector in a few selected vaccination centres located in the capital of Dhaka. Due to the limited availability of the vaccine in Bangladesh, the willingness to receive the influenza vaccine of risk group populations such as health care workers remains unclear.

To remedy this gap, this study intends to determine the current status of influenza vaccination among healthcare workers and generate preliminary data on whether increased awareness and availability of influenza vaccine improve vaccine uptake among healthcare workers and factors affecting the uptake rates. The critical data generated from the study would inform the development of an influenza vaccination policy among health care workers.

Research Design and Methods:

Study design:

The investigators will use a cluster randomized controlled trial design with the hospital as the unit of randomization and intervention. The intervention will be randomly allocated at the facility level and will include four arms: i) availability of influenza vaccine supply; ii) influenza vaccine awareness; iii) both influenza vaccine supply and influenza vaccine, and iv) control arm with no intervention. The investigators will assess influenza vaccine uptake before and after intervention and between different study arms. Moreover, barriers and motivators of vaccine uptake will be explored by applying a qualitative approach (i.e. in-depth interviews, key informant interviews, and focus group discussions). The investigators will also use a qualitative approach to understand the policy makers' perspectives and opinions on influenza vaccine uptake among HCWs.

Study site:

The study will be conducted at four purposively selected tertiary-level public teaching hospitals in Bangladesh. The investigators have chosen study hospitals considering several factors. Firstly, to minimize the diffusion of interventions, the investigators have selected hospitals from four different administrative divisions. Secondly, the investigators have avoided hospitals where the investigators have other ongoing studies among HCWs. Lastly, the investigators have chosen tertiary-level public hospitals with a higher number of HCWs to meet the minimum sample size requirement per study arm. The name and locations of the hospitals are as follows:

1. Sylhet MAG Osmani Medical College Hospital, Sylhet, Bangladesh
2. Rajshahi Medical College and Hospital, Medical College Road, Laxmipur, Rajpara, Rajshahi-6100, Bangladesh
3. Khulna Medical College Hospital, Sonadanga, Boyra, Khulna, Bangladesh
4. Mymensingh Medical College Hospital, Mymensingh, Bangladesh

Study population:

The study population would be HCWs, including doctors, nurses, and allied health personnel currently working at the study facilities. To ensure the support and co-operation of participating hospitals, the investigators will work closely with the participating hospital administration, including the hospital director. IEDCR will be our implementing partner for this project, and a letter of support from the director of IEDCR will be issued for all participating hospitals for their participation and co-operation. The investigators will collect the list of HCWs currently working in the facility from the hospital administration. The investigators will invite HCWs meeting our eligibility criteria to participate in the study.

Inclusion and exclusion criteria:

All HCWs who will be working at the study hospitals during the intervention period as well as consented to participate in the study will be included as participants.

HCWs not directly or indirectly involved in patient care, such as basic medical science faculties (e.g. anatomy, physiology, biochemistry, forensic medicine, pathology, and microbiology), will not be included as participants.

Intervention:

In Bangladesh, the Influenza season is between the late summer and rainy season, usually lasting from May to September. Before the start of the influenza season, the study hospitals will be randomly allocated into four study arms: 1) availability of influenza vaccine supply; 2) influenza vaccine awareness; 3) both influenza vaccine supply and influenza vaccine awareness, and 4) control arm with no intervention. The investigators will take the following measures for specific arms of intervention hospitals to inform study participants about receiving influenza vaccination.

Intervention arm-1: Intervention package with the availability of vaccine supply only

1.1. In Bangladesh, all vaccine suppliers currently sell inactivated, quadrivalent, and Northern Hemisphere flu vaccines. This vaccine contains influenza A(H3N2), pandemic A(H1N1), and influenza B lineage: B/Yamagata and B/Victoria. The investigators will work with the supplier to make that vaccine available at the hospital premises. Then a vaccination booth will be set up at the hospital premises and will administer the vaccine at the MRP.

1.2. All HCWs will be notified about only vaccine availability information by the hospital director and respective heads.

1.3. A list of all staff working in the study hospitals will be prepared, and they will be provided with an influenza vaccination record card with a unique identification number. The study staff will ensure receipt of vaccination cards for all participants.

1.4. No vaccine awareness information will be disseminated among the HCWs. 1.5. A short message (SMS) will be delivered over the mobile phone number to all participants, e.g. vaccination program duration, venue, time, and vaccine price, to cascade vaccination information to participants.

1.6. Posters with only vaccine delivery information (i.e. vaccination duration, vaccination venue, vaccine price) will be displayed at key hospital locations, e.g., the main entrance of the hospital, nursing station, vaccine delivery point/place, doctors' room, nurses' room, intern doctors' room, common room canteen etc.

Intervention arm-2: Intervention package with vaccination awareness only

2.1. The hospital director and respective heads will notify all HCWs about participating in the vaccination awareness program facilitated by the study team.

2.2. The investigators will arrange separate seminars for each group of HCWs (doctors, nurses, and allied health personnel) in the hospital to sensitize participants about the significance of receiving the influenza vaccine and the risk and benefits of influenza vaccination.

2.3. A list of all staff working in the study hospitals will be prepared, and they will be provided with an influenza vaccination record card with a unique identification number. The study staff will ensure receipt of vaccination cards for all participants.

2.5. A short message (SMS) will be delivered over the mobile phone number to all participants, e.g., time to vaccinate, vaccine price, and available places to purchase the vaccine.

2.6. Posters containing messages on the importance of influenza vaccination will be displayed at key hospital locations, e.g., the main entrance of the hospital, nursing station, vaccine delivery point/place, doctors' room, nurses' room, intern doctors' room, common room canteen etc.

2.4. No vaccination booth will be set up at the hospital premises.

Intervention arm-3: Intervention package with a combination of vaccine availability and awareness

3.1. The investigators will work with the study hospital authority, Influenza vaccine manufacturer, and supplier company to set up a vaccination booth at the hospital premises to administer the vaccine at the market-rated price (MRP) by hospital nurses.

3.2. The hospital director and respective department heads will notify all HCWs to receive the offered influenza vaccine.

3.3. A list of all staff working in the study hospitals will be prepared, and they will be provided with an influenza vaccination record card with a unique identification number. The icddr,b study staff will ensure receipt of vaccination cards for all participants.

3.4. The investigators will arrange separate seminars for each group of HCWs (doctors, nurses, and allied health personnel) in the hospital to sensitize participants about the objectives and implementation of the ongoing vaccination program as well as about the significance of receiving the influenza vaccine and the risk and benefits of influenza vaccination.

3.5. A short message (SMS) will be delivered over the mobile phone number to all participants, e.g. vaccination program duration, venue, time, vaccine price, to cascade vaccination information to optimum participants.

3.6. Posters with key messages will be displayed at key hospital locations, e.g., the main entrance of the hospital, nursing station, vaccine delivery point/place, doctors' room, nurses' room, intern doctors' room, common room canteen etc.

Control arm: No intervention

4.1. In the control facility, the investigators will not intervene in the existing knowledge and practice about influenza vaccination of the HCWs.

2. Implementing the vaccination program (for intervention arms 1 & 3)

A vaccination booth will be set up at the nurse's station or in a common space in both hospitals. The vaccine will be provided at MRP among HCWs. The hospital nurses will administer the vaccine. After receiving the vaccine, HCWs will sign the vaccination card in front of the staff nurse to ensure receiving a vaccine receipt. During the two-month vaccination program, icddr,b staff will monitor the entire program and ensure vaccine and logistics availability in study hospitals.

To report any adverse events following immunization (AEFI), the investigators will follow the existing surveillance channel established by the WHO and the Ministry of Health and Family Welfare (MoHFW), the government of Bangladesh. During the intervention briefing sessions at each study arm, the investigators will provide information about reporting an AEFI (if any) within the hospital's existing surveillance system as well as the hotline number (provided in the consent form) to inform such an issue. Moreover, throughout the study implementation period, an icddr,b staff will be placed at each study hospital, and he will also monitor any AEFI issue along with existing hospital surveillance set up. If any AEFI case is found, the icddr,b staff will immediately inform the Hospital Surveillance Officer (HSO), assist the HSO in filling in the AEFI report form, and submit it to the Expanded Programme on Immunization (EPI) headquarter through the Chief Health Officer. Besides, the investigators will analyse the AEFI data (i.e. the number of AEFI reports received, number of AEFI by type, and classification of AEFI by cause) and share the findings with key stakeholders, including the Directorate General of Drug Administration (DGDA).

Data collection:

1. Addressing Objective-1: To assess vaccine uptake The investigators will employ a quantitative method for evaluating vaccine uptake assessment. The investigators will perform the following activities- 1.1. The investigators will conduct a baseline survey among HCWs of the study facilities to collect information on influenza vaccine uptake history (have had ever and in the last influenza season) and knowledge status of influenza vaccine acceptance.

   1.2 At the end of the Influenza vaccine season, the investigators will do a post-intervention survey at study facilities to collect similar information.

   Trained staff will approach the participants to solicit their interest and consent. The staff will be well spoken and discuss with the study participants regarding confidentiality, objectives of the survey, use of data, and utility of results. Those who agree to participate will be interviewed according to the survey questionnaire. The structured questionnaire will be focused on the number of vaccinated HCWs (evidence from the signed vaccination card), socio-demographic information of the participants, including age, gender, profession (doctor/nurse), and department; perception of flu risk; perception of vaccine effectiveness and side effects, practices of recommending vaccination to family and patients, and practice and attitude towards a mandatory vaccination and their willingness to pay for future vaccination.
2. Addressing Objective-2: Understanding barriers and motivators for vaccination

   At the end of the intervention, both quantitative and qualitative surveys will be conducted to address objective 2. The quantitative survey will include structured questions on vaccine uptake motivators and barriers. Besides, qualitative methods (e.g., in-depth interviews (IDIs), focus group discussions (FGDs)) will be used to understand vaccinated and non-vaccinated participants' perceptions about influenza risk, vaccine effectiveness, side and adverse effects. The qualitative investigation will further effort to understand the experiences about the influenza vaccination i.e., barriers and motivators for vaccine acceptance. IDIs will be performed with both vaccinated and non-vaccinated HCWs to reveal an in-depth understanding of the factors and decisions for participating in vaccination. In addition, the investigators will carry out FGDs with intern doctors (to understand group behaviour and peer pressure on vaccination), nurses and allied health personnel for data triangulation and to comprehend the influence of group behaviour on vaccine uptake.

   For planning purposes, minimal sample sizes for each target group will be anticipated (Table 1) based on experiences from past studies. However, reduced or additional participants per target group may be recruited depending on the saturation point. Although an indicative minimal sample size has been provided (see list below), participants should be recruited until theoretical saturation for the research objective is reached, which is the point when no new insights are generated through the data

   Table-1: Distribution of IDIs and FGDs

   In-depth interviews (IDIs) participant selection (participants will be selected from years of experience, the domain of experience and male: female ratio will be maintained)

   Vaccinated-With doctors-4; Vaccinated-With nurses-4; Vaccinated-With allied health personnel-4; Non-vaccinated-With doctors-4; Non-vaccinated-With nurses-4; Non-vaccinated-With allied health personnel-4; Total number of IDI participants-24;

   Focus group discussions (heterogeneous in the combination of male-female participation; 8-10 participants in each discussion); Vaccinated-With doctors-1; Vaccinated-With nurses-1; Vaccinated-With allied health personnel-1; Non-vaccinated-With doctors-1; Non-vaccinated-With nurses-1; Non-vaccinated-With allied health personnel-1; Total number of FGDs-6;
3. Addressing Objective-3: Understanding the feasibility of influenza vaccination among HCWs To explore the feasibility of the influenza vaccination of HCWs, the investigators will carry out qualitative data collection by key-informant interviews (KIIs) with purposively selected personnel and stakeholders (Table 2). The qualitative data will be on experiences with influenza vaccination programs; barriers faced in implementing the vaccination program; existing workload; availability of infrastructural supports, logistics, and human resources; adequacy of cold chain and vaccine storage management; suitability of vaccination session management; and assessment of previous vaccination programs among health workers (if any), with particular attention to the feasibility of influenza vaccination among HCWs.

The investigators will conduct key informant interviews (KIIs) of the following key stakeholders (Table 2); however, the final number will depend on data saturation. The investigators will summarise the interview data to prepare a policy brief and share it with the NITAG.

Table-2: Distribution of KIIs Director, Communicable Disease Control, DGHS-1; Director, IEDCR, DGHS-1; Line Director, EPI-1; Program manager, EPI-1; Deputy program manager, EPI-1; Key personnel from WHO-1; Current and retired influenza experts-2; Members of the National Immunization Technical Advisory Group (NITAG)-2; GAVI Bangladesh-1; Hospital directors-4; Total number of interviews-15;

Sample Size Calculation:

This study's primary outcome of interest is influenza vaccine uptake among HCWs. An ongoing study among HCWs in Bangladesh at tertiary level facilities has shown an influenza vaccine uptake of about 5%. But Comprehensive reviews on influenza vaccine uptake among HCWs have shown a wide variation of vaccine uptake rates globally, between 13-53%. The investigators expect a similar uptake rate between 10-50% following awareness and availability of influenza vaccine supply in study hospitals. However, the investigators assume an increase in the uptake rate of at least five percentage points for the sample size requirement. With 80% power and a 5% level of significance, the investigators will require an estimated sample of size 435 HCWs in each arm to enroll in this study to detect a minimum increase of 5 percentage points in each intervention arm from the control arm of 5% expected uptake. With a clustering (design) effect of 2% and a 10% non-response rate, a sample size of 957 HCWs is required for each arm. Due to ethical considerations, the investigators plan to approach all healthcare workers (HCWs) in the study hospitals, which will result in an estimated total of 5759 healthcare workers, more than the estimated number of (957x4=3828); this would provide a more accurate estimate of the uptake rate and statistical power. An estimated number of HCWs in the study hospitals are given below.

Data Analysis:

The investigators will conduct a descriptive analysis to summarize the entire categorical variable using frequency, percentage, and 95% confidence interval. The investigators will summarize numerical or continuous variables using mean and standard deviation (SD) for symmetric distribution and median and interquartile range (IQR) for asymmetric distribution. The investigators will estimate the Difference in Differences (DID) with 95% CI of the proportion of vaccine uptake between each intervention and control (non-intervention) arm, adjusting for the clustering effect and testing whether it is statistically significant or not at a 5% level of significance. The investigators will also look for association and estimate the odds ratio (OR)/risk ratio (RR) with 95%CI between influenza vaccine uptake and its barriers and motivators, adjusting for clustering effect and covariates using multiple logistic regression/multilevel models.

For qualitative data, all the interviews will be transcribed verbatim in Bengali. Then the investigators will review some interviews to make initial code lists based on the interview guidelines and emerging themes for each group of respondents. After finalizing the code list, the team will code all the interviews and then summarize each code. Finally, the investigators will conduct a thematic analysis using a framework method.

Data Safety Monitoring Plan (DSMP):

This will not test any medical countermeasures. The intervention involves awareness and ensuring the availability of vaccine supply. The information collected from the respondents will be kept private, anonymous, and secret at all times. Participants' data privacy will be ensured, and all data collected throughout the research will be kept strictly confidential and won't be shared with anyone else. There will be no unauthorized access to this data. Also, there will be strong controls on who has access to the data forms and rigorous adherence to maintaining the data's confidentiality. There will be no sharing of participant names or any other identifying information with the information supplied by the survey respondents.

Ethical Assurance for Protection of Human rights:

The current protocol will determine the proportion of health care workers receiving influenza vaccines following awareness and availability of influenza vaccine supply. In addition, the study will also explore the factors associated with influenza vaccine uptake among healthcare workers.

This project will be based within hospital settings.

Sources of Material The staff will be well-spoken and discuss with the study participants regarding confidentiality, objectives of the survey, use of data, and utility of results. Those who agree to participate will be interviewed according to the survey questionnaire. All of the information will be recorded into a structured questionnaire electronically on TAB computers. The information of the participants will be recorded against a unique identification number. Only the study staff will have access to these records. The data will be entered into a password-protected computer.

Potential Risks This study poses minimal risk to participants from physical, psychological, financial, or legal perspectives. This project does not involve any therapeutic or novel interventions. The HCWs will be encouraged to take the influenza vaccine, which is safe and widely taken annually before the influenza season globally.

Recruitment and informed consent The study staff will approach the potential participant to inform him/her about the objectives of the study, study procedures, risks involved and invite him/her to participate. The participant will be enrolled in this study only after s/he has provided written informed consent.

Protection against risk The study physician will explain to participants the objectives, study procedures and risks involved in this study. The participant will be enrolled only after the provision of written informed consent. Risks to violation of confidentiality will be minimized, restricting access to the electronic database to everyone except the study staff. De-identified data will be prepared before sharing them with any researchers outside the circle of the study co-investigators.

Potential benefits The benefit to the participant through enrollment is that the participant will know about the importance of taking influenza vaccination, and those receiving vaccine will be protected from influenza illness, thereby reducing nosocomial influenza transmission. Data on the barriers and motivators of influenza vaccine uptake among healthcare workers would inform policy decisions to improve vaccine uptake among this high-priority group for influenza vaccination.

The risks are minimal, and the benefits are substantial. Thus, the activity does not burden the study subjects too onerous.

Importance of the knowledge to be gained This study would generate valuable data on the programmatic feasibility of HCWs' vaccination to observe the targeted influenza vaccination, HCWs' vaccine uptake, and factors associated with uptake rates. Through this assessment, constraints faced for providing vaccines, the capacity of the health facility, preparedness, and the presence of logistical equipment for implementing vaccination programs will be articulated. The findings from the study will inform policy decisions regarding influenza vaccination among HCWs.

Inclusion of women and minorities Participants will be enrolled based on their meeting the eligibility criteria. Sex/gender and racial/ethnic group will not be a criterion for enrolment.

Use of Animals:

No animals will be used for the study.

ELIGIBILITY:
Inclusion Criteria:

* All HCWs who will be working at the study hospitals during the intervention period as well as consented to participate in the study will be included as participants

Exclusion Criteria:

* HCWs not directly or indirectly involved in patient care, such as basic medical science faculties (e.g. anatomy, physiology, biochemistry, forensic medicine, pathology, and microbiology), will not be included as participants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-12-29 (Estimated); Study Completion 2023-02-12 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccine uptake among HCWs | up to 4 months
  The proportion of influenza vaccine uptake among health care workers before and after intervention and between different study arms

SECONDARY OUTCOMES:
Motivators and barriers of influenza vaccine uptake | up to 4 months
  Different motivators and barriers of influenza vaccine uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Sylhet MAG Osmani Medical College Hospital, Sylhet, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillari A, Polito F, Pucciarelli G, Serra N, Gargiulo G, Esposito MR, Botti S, Rea T, Simeone S. Influenza vaccination and healthcare workers: barriers and predisposing factors. Acta Biomed. 2021 Mar 25;92(S2):e2021004. doi: 10.23750/abm.v92iS2.11106. PMID 33855983
- [Background] Iuliano AD, Roguski KM, Chang HH, Muscatello DJ, Palekar R, Tempia S, Cohen C, Gran JM, Schanzer D, Cowling BJ, Wu P, Kyncl J, Ang LW, Park M, Redlberger-Fritz M, Yu H, Espenhain L, Krishnan A, Emukule G, van Asten L, Pereira da Silva S, Aungkulanon S, Buchholz U, Widdowson MA, Bresee JS; Global Seasonal Influenza-associated Mortality Collaborator Network. Estimates of global seasonal influenza-associated respiratory mortality: a modelling study. Lancet. 2018 Mar 31;391(10127):1285-1300. doi: 10.1016/S0140-6736(17)33293-2. Epub 2017 Dec 14. PMID 29248255
- [Background] Vanhems P, Benet T, Munier-Marion E. Nosocomial influenza: encouraging insights and future challenges. Curr Opin Infect Dis. 2016 Aug;29(4):366-72. doi: 10.1097/QCO.0000000000000287. PMID 27362641
- [Background] Lietz J, Westermann C, Nienhaus A, Schablon A. The Occupational Risk of Influenza A (H1N1) Infection among Healthcare Personnel during the 2009 Pandemic: A Systematic Review and Meta-Analysis of Observational Studies. PLoS One. 2016 Aug 31;11(8):e0162061. doi: 10.1371/journal.pone.0162061. eCollection 2016. PMID 27579923
- [Background] Kuster SP, Shah PS, Coleman BL, Lam PP, Tong A, Wormsbecker A, McGeer A. Incidence of influenza in healthy adults and healthcare workers: a systematic review and meta-analysis. PLoS One. 2011;6(10):e26239. doi: 10.1371/journal.pone.0026239. Epub 2011 Oct 18. PMID 22028840
- [Background] Apisarnthanarak A, Puthavathana P, Kitphati R, Auewarakul P, Mundy LM. Outbreaks of influenza A among nonvaccinated healthcare workers: implications for resource-limited settings. Infect Control Hosp Epidemiol. 2008 Aug;29(8):777-80. doi: 10.1086/588162. PMID 18624648
- [Background] Wilson KE, Wood SM, Schaecher KE, Cromwell KB, Godich J, Knapp MH, Sklar MJ, Ewing D, Raviprakash K, Defang G, Whitman TJ. Nosocomial outbreak of influenza A H3N2 in an inpatient oncology unit related to health care workers presenting to work while ill. Am J Infect Control. 2019 Jun;47(6):683-687. doi: 10.1016/j.ajic.2018.10.024. Epub 2019 Jan 5. PMID 30616930
- [Background] Chiu S, Black CL, Yue X, Greby SM, Laney AS, Campbell AP, de Perio MA. Working with influenza-like illness: Presenteeism among US health care personnel during the 2014-2015 influenza season. Am J Infect Control. 2017 Nov 1;45(11):1254-1258. doi: 10.1016/j.ajic.2017.04.008. Epub 2017 May 16. PMID 28526310
- [Background] Huttunen R, Syrjanen J. Healthcare workers as vectors of infectious diseases. Eur J Clin Microbiol Infect Dis. 2014 Sep;33(9):1477-88. doi: 10.1007/s10096-014-2119-6. Epub 2014 May 6. PMID 24798250
- [Background] Turnberg W, Daniell W, Duchin J. Influenza vaccination and sick leave practices and perceptions reported by health care workers in ambulatory care settings. Am J Infect Control. 2010 Aug;38(6):486-8. doi: 10.1016/j.ajic.2009.12.006. Epub 2010 Feb 21. PMID 20176412
- [Background] Barberis I, Myles P, Ault SK, Bragazzi NL, Martini M. History and evolution of influenza control through vaccination: from the first monovalent vaccine to universal vaccines. J Prev Med Hyg. 2016 Sep;57(3):E115-E120. PMID 27980374
- [Background] Gasparini R, Amicizia D, Lai PL, Bragazzi NL, Panatto D. Compounds with anti-influenza activity: present and future of strategies for the optimal treatment and management of influenza. Part II: Future compounds against influenza virus. J Prev Med Hyg. 2014 Dec;55(4):109-29. PMID 26137785
- [Background] Frenzel E, Chemaly RF, Ariza-Heredia E, Jiang Y, Shah DP, Thomas G, Graviss L, Raad I. Association of increased influenza vaccination in health care workers with a reduction in nosocomial influenza infections in cancer patients. Am J Infect Control. 2016 Sep 1;44(9):1016-21. doi: 10.1016/j.ajic.2016.03.024. Epub 2016 May 5. PMID 27158088
- [Background] Amodio E, Restivo V, Firenze A, Mammina C, Tramuto F, Vitale F. Can influenza vaccination coverage among healthcare workers influence the risk of nosocomial influenza-like illness in hospitalized patients? J Hosp Infect. 2014 Mar;86(3):182-7. doi: 10.1016/j.jhin.2014.01.005. Epub 2014 Feb 6. PMID 24581755
- [Background] Benet T, Regis C, Voirin N, Robert O, Lina B, Cronenberger S, Comte B, Coppere B, Vanhems P. Influenza vaccination of healthcare workers in acute-care hospitals: a case-control study of its effect on hospital-acquired influenza among patients. BMC Infect Dis. 2012 Feb 1;12:30. doi: 10.1186/1471-2334-12-30. PMID 22292886
- [Background] Vaccines against influenza WHO position paper - November 2012. Wkly Epidemiol Rec. 2012 Nov 23;87(47):461-76. No abstract available. English, French. PMID 23210147
- [Background] Al Awaidy S, Althaqafi A, Dbaibo G; Middle East/North Africa Influenza Stakeholder Network (MENA-ISN). A Snapshot of Influenza Surveillance, Vaccine Recommendations, and Vaccine Access, Drivers, and Barriers in Selected Middle Eastern and North African Countries. Oman Med J. 2018 Jul;33(4):283-290. doi: 10.5001/omj.2018.54. PMID 30038727
- [Background] Eaton JL, Mohr DC, McPhaul KM, Kaslow RA, Martinello RA. Access, Education and Policy Awareness: Predictors of Influenza Vaccine Acceptance Among VHA Healthcare Workers. Infect Control Hosp Epidemiol. 2017 Aug;38(8):970-975. doi: 10.1017/ice.2017.113. Epub 2017 Jun 23. PMID 28641586
- [Background] Abu-Gharbieh E, Fahmy S, Rasool BA, Khan S. Influenza vaccination: healthcare workers attitude in three Middle East countries. Int J Med Sci. 2010 Sep 21;7(5):319-25. doi: 10.7150/ijms.7.319. PMID 20922053
- [Background] Van Hooste WLC, Bekaert M. To Be or Not to Be Vaccinated? The Ethical Aspects of Influenza Vaccination among Healthcare Workers. Int J Environ Res Public Health. 2019 Oct 18;16(20):3981. doi: 10.3390/ijerph16203981. PMID 31635299
- [Background] Hollmeyer H, Hayden F, Mounts A, Buchholz U. Review: interventions to increase influenza vaccination among healthcare workers in hospitals. Influenza Other Respir Viruses. 2013 Jul;7(4):604-21. doi: 10.1111/irv.12002. Epub 2012 Sep 18. PMID 22984794
- [Background] Naleway AL, Henkle EM, Ball S, Bozeman S, Gaglani MJ, Kennedy ED, Thompson MG. Barriers and facilitators to influenza vaccination and vaccine coverage in a cohort of health care personnel. Am J Infect Control. 2014 Apr;42(4):371-5. doi: 10.1016/j.ajic.2013.11.003. PMID 24679562
- [Background] Thompson MG, Gaglani MJ, Naleway A, Ball S, Henkle EM, Sokolow LZ, Brennan B, Zhou H, Foster L, Black C, Kennedy ED, Bozeman S, Grohskopf LA, Shay DK. The expected emotional benefits of influenza vaccination strongly affect pre-season intentions and subsequent vaccination among healthcare personnel. Vaccine. 2012 May 21;30(24):3557-65. doi: 10.1016/j.vaccine.2012.03.062. Epub 2012 Apr 1. PMID 22475860
- [Background] Rashid H, Yin JK, Ward K, King C, Seale H, Booy R. Assessing Interventions To Improve Influenza Vaccine Uptake Among Health Care Workers. Health Aff (Millwood). 2016 Feb;35(2):284-92. doi: 10.1377/hlthaff.2015.1087. PMID 26858382
- [Background] Looijmans-van den Akker I, van Delden JJ, Verheij TJ, van der Sande MA, van Essen GA, Riphagen-Dalhuisen J, Hulscher ME, Hak E. Effects of a multi-faceted program to increase influenza vaccine uptake among health care workers in nursing homes: A cluster randomised controlled trial. Vaccine. 2010 Jul 12;28(31):5086-92. doi: 10.1016/j.vaccine.2010.05.003. Epub 2010 May 23. PMID 20580740
- [Background] Dini G, Toletone A, Sticchi L, Orsi A, Bragazzi NL, Durando P. Influenza vaccination in healthcare workers: A comprehensive critical appraisal of the literature. Hum Vaccin Immunother. 2018 Mar 4;14(3):772-789. doi: 10.1080/21645515.2017.1348442. Epub 2017 Oct 20. PMID 28787234
- [Background] Azziz-Baumgartner E, Alamgir AS, Rahman M, Homaira N, Sohel BM, Sharker MA, Zaman RU, Dee J, Gurley ES, Al Mamun A, Mah-E-Muneer S, Fry AM, Widdowson MA, Bresee J, Lindstrom S, Azim T, Brooks A, Podder G, Hossain MJ, Rahman M, Luby SP. Incidence of influenza-like illness and severe acute respiratory infection during three influenza seasons in Bangladesh, 2008-2010. Bull World Health Organ. 2012 Jan 1;90(1):12-9. doi: 10.2471/BLT.11.090209. Epub 2011 Oct 4. PMID 22271960
- [Derived] Hassan MZ, Shirin T, Rahman M, Alamgir ASM, Jahan N, Al Jubayer Biswas MA, Khan SH, Basher MAK, Islam MA, Hussain K, Islam MN, Rabbany MA, Haque MA, Chakraborty SR, Parvin SR, Rahman M, Chowdhury F. Seasonal influenza vaccine uptake among healthcare workers in tertiary care hospitals, Bangladesh: Study protocol for influenza vaccine supply and awareness intervention. BMC Public Health. 2022 Sep 24;22(1):1819. doi: 10.1186/s12889-022-14182-w. PMID 36153529
- See also: WHO seasonal influenza vaccination recommendations during the COVID-19 pandemic - Recommandations du SAGE de l'OMS pour la vaccination contre la grippe saisonnière pendant la pandémie de COVID-19 — https://apps.who.int/iris/handle/10665/336260
- See also: Seasonal influenza vaccine use in low and middle income countries in the tropics and subtropics: a systematic review — https://apps.who.int/iris/handle/10665/188785
- See also: Health conditions for travellers to Saudi Arabia Pilgrimage to Mecca (Hajj) = Dispositions sanitaires pour les voyageurs se rendant en Arabie saoudite Pèlerinage à La Mecque (Hadj) — https://apps.who.int/iris/handle/10665/232956
- See also: Global Influenza Strategy 2019-2030 — https://www.who.int/publications-detail-redirect/9789241515320